CLINICAL TRIAL: NCT02405247
Title: TAURAS - T790 AURA ScreenFailure SOC Registry Study
Acronym: TAURAS
Status: Terminated | Type: Observational
Why Stopped: Team's request.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00003
Record Dates: First submitted 2015-03-16; First posted 2015-04-01 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; T790M; EGFR; TKI; Resistance; Non Small Cell Lung Cancer; AZD9291
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NSCLC without T790M mutation: NSCLC patients who have failed first line TKI treatment (defined radiological documentation of disease progression during treatment for advanced or metastatic NSCLC with an approved EGFR-TKI e.g. gefitinib, afatinib or erlotinib) and are screened for the AURA3 study and determined to be lacking the T790M mutation as determined using the AURA3 designated central laboratory using the cobas® EGFR Mutation Test (Roche Molecular Systems).
  Interventions: Other: Patient Reported Outcome (PRO)

INTERVENTIONS:
Other: Patient Reported Outcome (PRO) — Exposure to Quality of Life Questionnaires (EORTC QLQ-LC13, EORTC QLQ-C30 and EQ-5D-5L) every 3 months during standard of care visits.

SUMMARY:
The aim of this study is to evaluate clinical outcomes of 2nd line therapy in NSCLC patients without the T790M mutation, both independently and when compared indirectly with NSCLC patients with the T790M mutation in the T STAR non interventional study (D5160R00001).

The patient population in the TAURAS study will consist of patients who fail screening for AURA3 (D5160C00003) due to a T790M mutation not detected using the central cobas® EGFR Mutation Test (Roche Molecular Systems).

DETAILED DESCRIPTION:
The study design is an observational prospective cohort study. The study plans to enroll approximately 400 patients from an estimated 17 countries.

Patients will be recruited from the patient pool that is being screened for the AZD9291 AURA3 randomized clinical trial (RCT). Biopsy tissues and consents have already been obtained from patients to use samples for future research as part of the AURA3 trial screening processes. During the RCT screening process, the patients sign a full consent to participate in the AURA3 trial, and have their tumour tested as part of the main screening.

Data are collected, notably on medical history, co-medications, and adverse events. Biopsy tissue is collected to assess T790M mutation status. All patients will be able to enter the TAURAS study regardless of whether or not they have any remaining tissue. Biomarker analyses resulting from the historical tumour samples obtained as part of the AURA3 screening process, and in accordance with the consent obtained within the AURA3 trial protocol, can be linked to the data collected in TAURAS and used as part of the exploratory objectives of this NIS.

The primary objectives of the NIS study in NSCLC patients who have progressed on a previous EGFR-TKI (with no intervening chemotherapy) and who do not harbour the T790M mutation (according to central analysis using the Roche cobas® EGFR Mutation Test), are:

* To estimate overall survival
* To estimate disease progression (as assessed and defined by physician)
* To estimate partial, complete, and overall response rates by line of therapy (as assessed and defined by physician)
* To describe treatment patterns for 2nd line and beyond, including time on treatment by line of therapy and time to subsequent therapies (or death)
* To describe health resource utilization patterns (e.g., hospitalizations, emergency room visits)
* To capture patient reported symptoms, functioning and health-related quality of life (HRQoL) data using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30), and European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13)
* To capture health state utilities using the EQ-5D-5L questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent from the patient or next-of-kin for deceased patient at study entry, where this is mandated/allowed by local regulations
2. Aged at least 18 years. Patients from Japan aged at least 20 years
3. Patients who have been considered ineligible for entry into the AZD9291 AURA3 registration trial as a result of their tumour not harbouring the T790M mutation, according to the cobas EGFR test of a biopsy taken following the latest line of therapy, at a central testing lab participating in the D5160C00003 (AURA3) study.
4. Patients who have undertaken or plan to undertake 2nd-line therapy after screen failure for the AURA3 study.

Exclusion Criteria:

1. Treatment with any of the following:

   * Prior treatment with more than one line of systemic treatment for advanced disease prior to failing screening assessments for AURA3.
   * Major surgery (excluding placement of vascular access) within 4 weeks prior to failing screening assessments for AURA3.
   * Palliative radiotherapy with a limited field of radiation within 1 week prior to enrolment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks prior to failing screening assessments for AURA3..
2. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to failing screening assessments for AURA3..
3. Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the study site).
4. Judgment by the physician that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
5. Patients who are known to be entering an interventional clinical study (blinded, randomized or open label clinical study) at the time of the enrolment into this study. However, inclusion in this study does not preclude participation in any other clinical study after enrolment. Patients who participate in clinical studies after enrolment into this study will be followed up to the extent possible as permitted by the sponsor of that clinical study.
6. Patients with an invalid or unsuccessful T790M mutation test result during screening for AURA3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients who have failed first line TKI treatment (defined radiological documentation of disease progression during treatment for advanced or metastatic NSCLC with an approved EGFR-TKI e.g. gefitinib, afatinib or erlotinib) and are screened for the AURA3 study and determined to be lacking the T790M mutation as determined using the AURA3 designated central laboratory using the cobas® EGFR Mutation Test (Roche Molecular Systems). Only sites that are participating in the AURA3 study, and patients who had the T790M mutation tested for AURA3 screening (and determined not to have the T790M mutation) will be included.
  The study plans to enroll approximately 400 patients from approximately 136 sites in an estimated 17 countries globally.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 24 months from last subject in
  This will be assessed as the time from start of 2nd line therapy until the date of disease progression or death by any cause.
Response to Therapy as assessed by the physician | 24 months from last subject in
  This will be assessed as the time from start of 2nd line therapy until the date of disease progression or death (by any cause in the absence of progression). To assess efficacy of 2nd line treatment and beyond.
Time on treatment by line of therapy and between therapies | 24 months from last subject in
  This will be assessed as the time from start date of line of therapy to end date of line of therapy or death date. To describe treatment patterns for 2nd line and beyond.
Admission of planned/unplanned hospitalizations, emergency department visits and outpatient/physician visit | 24 months from last subject in
  This will be assessed as the number and Time from the dates of admission and exit of attendance. To describe Healthcare resource utilization for 2nd line treatment and beyond.
Time to symptom deterioration | 24 months from last subject in
  For each of the symptoms in EORTC QLQ-LC13 and EORTC QLQ-C30, Time from inclusion until the date of first clinically meaningful symptom deterioration or death by any cause in the absence of a clinically meaningful symptom deterioration. To assess the impact of 2nd and subsequent lines of therapy on patients' disease-related symptoms and health related quality of life.
Symptom Improvement Rate | 24 months from last subject in
  This will be assessed as the number of patients with two consecutive assessments, which showed a clinically meaningful improvement in that symptom from baseline. To assess the impact of 2nd and subsequent lines of therapies on patients' disease-related symptoms and health related quality of life.
Overall Survival | 24 months from last subject in
  This will be assessed as the time from the start date of 2nd line chemotherapy until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Research Site, Oceanside, California
  - Research Site, Santa Rosa, California
- South Korea (3):
  - Research Site, Seongnam, Gyeonggido
  - Research Site, JinJoo, Gyeongsangnam-do
  - Research Site, Ulsan, Ulsan Gwangyeogsi